CLINICAL TRIAL: NCT00497016
Title: Does Statin Therapy Reduce Sympathoexcitation in Hypertension?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: HTSTAT
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Hypertension
Keywords: hypertension; statin; sympathetic
MeSH Terms: conditions — Hypertension | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin 80 mg

SUMMARY:
A number of patients with hypertension have increased central sympathetic activity. Statins seem to inhibit central sympathetic output. This study assesses the effect of statins on central sympathetic activity in hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* (Known) hypertension
* stable drug therapy for at least 2 months
* age 18-70 jaar
* BMI 18-35 kg/m2
* Sinusrhythm

Exclusion Criteria:

* Recent cardiovascular event <6 mnd
* Plasma Creatinin:
* female: >120 mmol/L
* male: >133 mmol/L
* use of:
* tricyclic antidepressants
* alpha-1 -and/or alpha-2 blockers
* disease of the autonomic nervous system (Parkinsons disease, Shy- Drager syndrome, etc)
* Albuminuria >300 mg/dag

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2007-05; Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
change in central sympathetic activity

SECONDARY OUTCOMES:
change in cholesterol levels, renin and aldosteron

CONTACTS AND LOCATIONS:
Overall Officials: Cees J Tack, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Center Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Derived] Gomes ME, Tack CJ, Verheugt FW, Smits P, Lenders JW. Sympathoinhibition by atorvastatin in hypertensive patients. Circ J. 2010 Nov;74(12):2622-6. doi: 10.1253/circj.cj-10-0427. Epub 2010 Oct 9. PMID 20953062